CLINICAL TRIAL: NCT06948539
Title: A Phase I Clinical Trial Evaluating the Tolerability and Pharmacokinetics of TQB2101 for Injection in Subjects With Advanced Malignancies
Brief Title: To Evaluate the Tolerability and Pharmacokinetics of TQB2101 for Injection in Patients With Advanced Malignant Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2101-I-01
Record Dates: First submitted 2025-04-17; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Lung Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2101 injection (Experimental): The drug was administered every 3 weeks for 21 consecutive days in a treatment cycle.
  Interventions: Drug: TQB2101 for injection

INTERVENTIONS:
Drug: TQB2101 for injection — TQB2101 for injection is a receptor tyrosine kinase-like orphan receptor-1 antibody drug conjugate.

SUMMARY:
To explore the tolerability and pharmacokinetics of TQB2101 for injection in subjects with advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and had good compliance;
* 18 years old ≤ age ≤75 years old (calculated on the date of signing the informed consent);
* Eastern Cooperative Oncology Group (ECOG) score 0~1;
* Expected survival greater than 12 weeks;
* Patients with advanced solid tumors confirmed by cytology/histopathology, failure of standard treatment or lack of effective treatment ; Participants with Receptor Tyrosine Kinase-Like Orphan Receptor 1 (ROR1) -positive advanced solid tumors were enrolled in the extended study phase.
* Evidence of at least one measurable lesion according to RECIST 1.1 criteria, except that the dose-escalation phase is not required to be measurable, as long as it meets the assessment of disease status.
* The main organs function well and meet the following criteria:

  1. Hemoglobin (HGB) ≥80g/L;
  2. Absolute neutrophil count (ANC) of solid tumor subjects ≥1.5×109 /L;
  3. Platelet count (PLT) ≥100×109/L, if accompanied by bone marrow invasion, platelet ≥75×109/L;
  4. Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN);
  5. Alanine transferase (ALT) and aspartate transferase (AST) ≤2.5×ULN. ALT and AST≤5×ULN if accompanied by liver metastasis;
  6. Serum creatinine (CR) ≤1.5×ULN or creatinine clearance (CCR) ≥60 mL /min (standard Cockcroft-Gault formula was applied;
  7. Prothrombin time (PT), activated partial thromboplastin time (APTT), International standardized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy);
* Women of reproductive age should agree that effective contraception must be used during the study period and for 6 months after the end of the study, and that serum or urine pregnancy tests are negative within 7 days prior to study enrollment; Men should agree that effective birth control must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Had or was currently suffering from other malignant tumors within 3 years prior to the first medication.
* There are multiple factors that affect intravenous injection, venous blood collection diseases, or have an impact on oral drugs.
* The adverse reactions of previous treatment failed to recover to Common Terminology Criteria for Adverse Events Version 5 (CTCAEv5.0) score ≤1.
* Patients who had major surgical treatment, significant traumatic injury, or potential major surgery during the expected study treatment period within 4 weeks prior to initial medication, or who had long-term unhealed wounds or fractures.
* Subjects who have had any bleeding event ≥CTCAEv5.0 level 3 within 4 weeks prior to initial dosing, or who have bleeding or clotting disease and are taking warfarin, aspirin, or other antiplatelet agglutinating agents (except maintenance doses) : Subjects with aspirin ≤100mg/ day, clopidogrel ≤75mg/ day, or with any signs of bleeding or medical history determined by the investigator to be unsuitable for enrollment.
* Patients who experienced a hyperarterial/venous thrombosis event, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, within 6 months before the first administration of the drug.
* Chronic hepatitis B active or active hepatitis C subjects. Subjects who are positive for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies during screening should undergo Hepatitis B Virus (HBV) DNA titer testing or HCV RNA testing.
* Patients with active syphilis who need treatment.
* There is a history of active pulmonary tuberculosis, idiopathic pulmonary fibrosis, institutional pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment, or active pneumonia with clinical symptoms.
* Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders.
* Decompensated stage of cirrhosis and history of hepatic encephalopathy.
* Subjects with clinically significant cardiovascular disease, including any of the following:

  1. Participants who had acute myocardial infarction and severe/unstable angina pectoris within 6 months before the start of study treatment; Or have heart failure of the New York Heart Association's heart function classification level 2 or higher;
  2. QT interval prolongation at rest as corrected by Fridericia Formula (QTcF), QTc interval ≥450ms(male), QTc interval ≥470 ms(female);
  3. Have a past or ongoing history of severe uncontrolled ventricular arrhythmias requiring medical treatment;
  4. Left ventricular ejection fraction (LVEF) < 50%;
  5. Congenital long QT syndrome, or any known history of tip torsion ventricular Torsades de Pointes (TdP);
  6. Clinically uncontrolled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg after standard antihypertensive therapy) and a history of hypertensive encephalopathy/hypertensive crisis.

Active or uncontrolled severe infection (≥CTC AEv5.0 grade 2 infection).

* Patients with renal failure requiring hemodialysis or peritoneal dialysis.
* Have a history of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases.
* Subjects with (non-infectious) pneumonia/interstitial lung disease requiring steroid treatment or who currently have non-infectious pneumonia/interstitial lung disease or have been hospitalized for any active infection or received therapeutic antibiotics in the 4 weeks prior to beginning study treatment, including but not limited to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection.
* People who have epilepsy and need treatment.
* Urine routine indicated urine protein ≥ ++, and confirmed 24-hour urine protein quantity > 1.0 g.
* Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L).
* Tumor-related symptoms and treatment:

  1. For subjects who have received chemotherapy, immunotherapy within 4 weeks prior to the first dose, radiation therapy or small molecule targeted drugs within 2 weeks, or who are still within the 5 half-lives of the drug (depending on the shortest time of occurrence), the washout period is calculated from the end time of the last treatment;
  2. Within 2 weeks before the first drug use, it has been treated with Chinese patent medicines (including compound Cantharides capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Bruceae oil injection/capsule, Xiaoaiping tablet/injection, hualbufatin capsule, etc.) with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions;
  3. Imaging (CT or MRI) shows that the tumor has invaded important blood vessels, or the investigator determines that the tumor is highly likely to invade important blood vessels during the follow-up study period and cause fatal massive bleeding;
  4. Uncontrolled pleuroceliac or pericardial effusion requiring repeated drainage or obvious symptoms. Subjects who are asymptomatic and have not received drainage or other treatment in the first 2 weeks of enrollment can be enrolled if imaging shows only small amounts of pleural effusion, ascites, or pericardial effusion.
* Known allergy to study drug excipients.
* Previous therapy with targeted ROR1 inhibitors.
* Participants who have participated in a clinical trial of another antitumor drug (calculated as the last use of the investigational drug) within 4 weeks prior to initial administration and have used the investigational drug, or are still within 5 half-lives of the investigational drug (whichever is shorter).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase II recommended doses (RP2D) | Baseline up to 24 months
  The dosage of drug therapy recommended for use in the second phase of clinical trials (i.e., phase II clinical trials).
Dose-limiting toxicity (DLT) | Up to 1 month
  Adverse events that meet the protocol definition of dose-limiting toxic event timing were evaluated according to the Common Terminology Criteria for Adverse Events 5.0.
Maximum tolerated dose (MTD) | Up to 1 month
  The previous dose of the dose group in which dose-limiting toxicity occurs is the maximum tolerated dose.

SECONDARY OUTCOMES:
Incidence and severity of adverse event (AE) and serious adverse event (SAE), and abnormal laboratory test indicators | Up to 24 months
  Incidence and severity of AE and SAE, and abnormal laboratory test indicators
Peak time | Up to 4 months
  Time to peak blood concentration after a single dose.
Peak concentration Cmax | Up to 4 months
  After a single dose, the highest point of the drug-time curve is called the peak concentration.
Plasma elimination half-life t1/2 | Up to 4 months
  The amount of time it takes for the concentration of the drug in the blood, or the amount of drug in the body, to drop to about half of its original level.
Objective response rate | Up to 24 months
  The objective response rate of injection form TQB2101 in patients with advanced solid tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Prevention Center, Guanzhou, Guangdong, China